CLINICAL TRIAL: NCT03087422
Title: An Intervention Based on Text Message (SMS) to Help Cancer Patients in Chemotherapy Treatment
Brief Title: Text Message (SMS) to Help Cancer Patients in Chemotherapy Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samanta Winck Madruga (Other)
Responsible Party: Sponsor-Investigator, Samanta Winck Madruga, Hospital Escola, Federal University of Pelotas
Organization: Federal University of Pelotas (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HospitalEscolaUFPel
Record Dates: First submitted 2017-03-03; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Cancer; Side Effect
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): The patients in this group will receive daily a text message (SMS) with some orientation about Homecare as an attempt to minimize the side effects of chemotherapy.
  The text messages are based on oncology guidelines.The text messages contain information about water intake, emotional support, hygiene, immunity, nutrition, and physical activity. In addition, text messages about prevention and management of symptoms were also developed: nausea and vomiting, diarrhea, constipation, gas, changes in the skin and taste.
  Also, the patients allocated in this group will receive the standard care.
  Interventions: Behavioral: Text message intervention
- control (No Intervention): The patients allocated in this group will receive the standard care.

INTERVENTIONS:
Behavioral: Text message intervention — The intervention consists in sending text messages with orientation that helps in homecare, specifically attempting to minimize chemotherapy side effects.
  Arms: intervention

SUMMARY:
This study evaluates the text message (SMS) with orientation to help the management of chemotherapy treatment.

DETAILED DESCRIPTION:
The investigators developed an app (called ChemotherApp) for Android that automatically sends text messages with homecare orientation to cancer patients in intervention group. The main features of this app are: to register information such as name, number of cellphone, gender, and chemotherapy schedule of the patient. Other feature is to register the orientation that will be sent to patients by text messages. Daily, the app send a registered orientation to each patient.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients who will start chemotherapy treatment in Hospital Escola of Federal University of Pelotas.

Exclusion Criteria:

* Illiterate patients; Patients who do not have their own cell phone

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-12-15 (Estimated)

PRIMARY OUTCOMES:
Change from Chemotherapy Side Effects - QLQ-C30 EORTC questionnaire | Up to 4 month
  To measure the side effects, the QLQ-C30 EORTC questionnaire is going to be used. This questionnaire aims to identify if the patient had nausea and vomit, diarrhea, pain, fever, constipation, diarrhea, gas, among other symptoms. It will be investigated if patients who will receive the text message will have less side effects than patients who will not receive text messages. The questionnaire will be applied to each patient in the study at the beginning of the second,third and fourth cycles of chemotherapy.

SECONDARY OUTCOMES:
Change from Anxiety and Depression - HADS (Hospital Anxiety and Depression Scale) questionnaire | Up to 4 month
  To measure anxiety and depression, the HADS (Hospital Anxiety and Depression Scale) questionnaire is going to be used. It will be investigated if patients who will receive the text message will have less score of depression and anxiety than patients who will not receive text messages. The HADS questionnaire is going to be applied to each patient on the first day of treatment and at the beginning of the fourth cycle of chemotherapy.

OTHER OUTCOMES:
Change from ECOG (The Eastern Cooperative Oncology Group) scale - performance status - well-being | Up to 4 month
  ECOG (The Eastern Cooperative Oncology Group) scale will be used to evaluate the performance status,to measure the well-being. It will be investigated if patients who will receive the text message will have better performance status than patients who will not receive text messages. A performance status will be evaluated at the beginning of treatment and at the beginning of the second cycle of chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rico TM, Dos Santos Machado K, Fernandes VP, Madruga SW, Santin MM, Petrarca CR, Dumith SC. Use of Text Messaging (SMS) for the Management of Side Effects in Cancer Patients Undergoing Chemotherapy Treatment: a Randomized Controlled Trial. J Med Syst. 2020 Sep 30;44(11):193. doi: 10.1007/s10916-020-01663-x. PMID 32996027